CLINICAL TRIAL: NCT04983641
Title: Pre-visit Digital Messaging Improves Patient Reported Outcome Measure Participation Prior to the Orthopedic Ambulatory Visit: A Prospective, Randomized, Control Trial
Brief Title: Pre-visit Digital Messaging Improves Patient Reported Outcome Measure Participation Prior to the Orthopedic Ambulatory Visit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Eric Makhni, Medical Director, Center for Patient Reported Outcome Measures; Director of Quality and Informatics, Orthopedic Service Line, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 13895
Record Dates: First submitted 2021-07-03; First posted 2021-07-30 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Orthopedic Disorder
Keywords: PROMIS; Patient Reported Outcomes Measurement Information System
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control - No Pre-Visit Message (No Intervention): o Patients were assigned PROMIS forms in the domains of Depression (PROMIS-D) and Pain Interference (PROMIS-PI) in addition to Upper Extremity Function (PROMIS-UE) and/or Physical Function (PROMIS-PF). These forms were available for remote completion in each respective patient's MyChart portal at 1 week prior to their clinic appointment. Patients in this arm were not sent any reminder e-mails or MyChart messages concerning PROMIS form completion at any timepoint prior to their scheduled clinic visit.
- E-mail Arm (Experimental): o Patients were assigned PROMIS forms in the domains of Depression (PROMIS-D) and Pain Interference (PROMIS-PI) in addition to Upper Extremity Function (PROMIS-UE) and/or Physical Function (PROMIS-PF). These forms were available for remote completion in each respective patient's MyChart portal at 1 week prior to their clinic appointment. Patients in this arm were sent an initial reminder e-mail message at 1 week prior to their scheduled clinic visit regarding PROMIS form completion. If patient's did not fill out PROMIS forms by 3 days prior to their visit, they were sent a second reminder e-mail message.
  Interventions: Other: Pre-Visit Messages
- Digital Patient Portal "MyChart" Arm (Experimental): o Patients were assigned PROMIS forms in the domains of Depression (PROMIS-D) and Pain Interference (PROMIS-PI) in addition to Upper Extremity Function (PROMIS-UE) and/or Physical Function (PROMIS-PF). These forms were available for remote completion in each respective patient's MyChart portal at 1 week prior to their clinic appointment. Patient's in this arm were sent an initial reminder MyChart message at 1 week prior to their scheduled clinic visit regarding PROMIS form completion. If patients did not fill out PROMIS forms by 3 days prior to their visit, they were sent a second reminder MyChart message.
  Interventions: Other: Pre-Visit Messages

INTERVENTIONS:
Other: Pre-Visit Messages — Patients in both experimental arms (E-mail and Digital Patient Portal "MyChart") were sent pre-visit messages regarding PROMIS form completion via each respective modality at 1 week and also 3 days prior to their respective Orthopaedic clinic visits
  Arms: Digital Patient Portal "MyChart" Arm; E-mail Arm

SUMMARY:
Patient-Reported Outcomes Measurement Information System (PROMIS) forms will be administered remotely to consecutive Orthopaedic patients presenting for new physician clinic visits. These patients will be sent either reminder e-mails, reminder digital patient portal ("MyChart") messages, or no reminder messages at all concerning PROMIS form completion at timepoints prior to their respective clinic visits and PROMIS form completion rates will consequently be assessed. The primary objective of this study is to develop an understanding of whether pre-visit reminder messages influence PROMIS form completion in Orthopaedic patients.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* English speaking
* No previous PROM form completion at the healthcare system
* Seeing a respective orthopedic provider for the first time
* Active registration with the electronic medical record (EMR; Epic, Verona, WI) patient portal ("MyChart")
* Valid e-mail address.

Exclusion Criteria:

* Under 18 years old
* Non-English speaking
* Previous PROM form completion at the healthcare system
* Seeing a respective orthopedic provider for follow-up
* No active registration with the electronic medical record (EMR; Epic, Verona, WI) patient portal ("MyChart")
* No valid e-mail address.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 291 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-12-07 (Actual); Study Completion 2020-12-07 (Actual)

PRIMARY OUTCOMES:
Pre-visit PROMIS completion rates in orthopaedic patients receiving reminder e-mails, digital patient portal ("MyChart") message reminders, or no messages prior to scheduled clinic visit | 1 week
  Investigators will assess whether reminder messages prior to clinic visit have an impact on both remote pre-visit and overall PROMIS form completion rates in orthopaedic patients. Patients completing a single assigned PROMIS form will be regarded as having PROMIS completion.
At-visit PROMIS completion rates in orthopaedic patients receiving reminder e-mails, digital patient portal ("MyChart") message reminders, or no messages prior to scheduled clinic visit | 1 week
  Investigators will assess whether reminder messages prior to clinic visit have an impact on both remote pre-visit and overall PROMIS form completion rates in orthopaedic patients. Patients completing a single assigned PROMIS form will be regarded as having PROMIS completion.
Overall (Pre-visit and at-visit) PROMIS completion rates in orthopaedic patients receiving reminder e-mails, digital patient portal ("MyChart") message reminders, or no messages prior to scheduled clinic visit | 1 week
  Investigators will assess whether reminder messages prior to clinic visit have an impact on both remote pre-visit and overall PROMIS form completion rates in orthopaedic patients. Patients completing a single assigned PROMIS form will be regarded as having PROMIS completion.

SECONDARY OUTCOMES:
Time to pre-visit PROMIS form completion | 1 week
  This is achieved by assessing the timepoint (in days) at which patients completed assigned PROMIS forms prior to their respective clinic visit in each of the designated study arms.
PROMIS form completion rates according to patient demographics | 1 week
  This is achieved by assessing how PROMIS form completion for the enrolled study cohort as a whole (irrespective of arm assignment) varies according to patient race, age, gender, and sub-specialty of visit

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
We are not sharing individual participant data.